CLINICAL TRIAL: NCT03974074
Title: Albumin Infusion for Patients With Hepatocellular Carcinoma and Hypoproteinemia After Hepatectomy
Brief Title: Albumin for Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Principal Investigator, Guangxi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Alb-HCC
Record Dates: First submitted 2019-05-30; First posted 2019-06-04 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hepatocellular Carcinoma; Hypoproteinemia
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypoproteinemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin infusion group (Experimental): Albumin infusion (20 g, ivgtt, qd) will be performed to patients with HCC after hepatic resection in 24 h for three days. All patients wil receive furosemide (10 mg, iv) after albumin transfusion. In the fifth day after resection, patients will receive albumin transfusion if they have ascites with shifting dullness, moderate edema (below both lower ankle joints) with serum albumin lower than 30 g/L, severe postoperation complication (septicopyemia, postoperative bleeding with reoperation, or biliary fistula).
  Interventions: Drug: Albumin infusion
- Empty control (No Intervention): Conventional liver protection and rehydration therapy.In the fifth day after resection, patients will receive albumin transfusion if they have ascites with shifting dullness, moderate edema (below both lower ankle joints) with serum albumin lower than 30 g/L, severe postoperation complication (septicopyemia, postoperative bleeding with reoperation, or biliary fistula).

INTERVENTIONS:
Drug: Albumin infusion — Albumin infusion (20 g, ivgtt, qd) will be performed to patients with HCC after resection in 24 h for three days.
  Arms: Albumin infusion group

SUMMARY:
The rate of liver cirrhosis is about 40% to 75% among patients with hepatocellular carcinoma (HCC). Therefore, many patients with HCC were with low serum albumin before and after (especially) hepatic resection. Serum albumin level has been routinely used in clinical practice as a surrogate marker to evaluate nutritional status and liver function. Serum albumin concentration is used as an independent mortality risk predictor in a broad range of clinical and research settings. However, the role of albumin infusion in patients with hepatocellular carcinoma (HCC) after resection is unknown. The present study aimed to investigate the safety and clinical necessity of albumin infusion for HCC patients after hepatic resection.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >18.5;
* Patients with primary hepatocellular carcinoma without any treatments for tumors before resection;
* Hepatocellular carcinoma should be confirmed by histopathology;
* With preserved liver function (Child-Pugh score ≤7) before resection
* ECOG performance score 0 or 1;
* Preoperative serum albumin >35g/L;
* The level of postoperative serum albumin is between 25-30g/L in the first day after resection.

Exclusion Criteria:

* Patients used albumin before liver resection (<1 months);
* Plasma was used during or after liver resection;
* Surgery involving the extrahepatic bile duct or gastrointestinal tract.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum total bilirubin level | Change from Baseline total bilirubin at the fifth and seventh days after resection
  Recovery of liver function between the two groups
Serum albumin level | Change from Baseline serum albumin at the fifth and seventh days after resection
  Recovery of liver function between the two groups

SECONDARY OUTCOMES:
Abdominal girth | Change from Baseline abdominal girth at the fifth and seventh days after resection
  Drainage liquid and abdominal girth between the two groups were compared
Rate of postoperative complications | The first months after resection
  The rate of postoperative complications between the two groups were compared

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Zhong Tang, MD, Study Director — Cancer Hospital of Guangxi Medical University
Locations (2):
- China (2):
  - Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Jian-Hong Zhong, Nanning, Guangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Result] Pericleous M, Sarnowski A, Moore A, Fijten R, Zaman M. The clinical management of abdominal ascites, spontaneous bacterial peritonitis and hepatorenal syndrome: a review of current guidelines and recommendations. Eur J Gastroenterol Hepatol. 2016 Mar;28(3):e10-8. doi: 10.1097/MEG.0000000000000548. PMID 26671516